CLINICAL TRIAL: NCT00778583
Title: An Open Label, Randomised, Two-Treatment, Four-Period, Two-Sequence, Single-Dose, Crossover, Fully Replicated Bioavailability Study on Nitrofurantoin Formulations Comparing Nitrofurantoin 100 mg Capsules of Ranbaxy Laboratories With Macrobid 100 mg Capsules in Healthy, Adult, Human Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Nitrofurantoin 100 mg Capsules Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 024/NITRO-100/03
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Nitrofurantoin capsules
MeSH Terms: interventions — Nitrofurantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Nitrofurantoin 100 mg capsules of Ranbaxy
  Interventions: Drug: Nitrofurantoin 100 mg capsules
- 2 (Active Comparator): Macrobid 100 mg capsules
  Interventions: Drug: Nitrofurantoin 100 mg capsules

INTERVENTIONS:
Drug: Nitrofurantoin 100 mg capsules

SUMMARY:
An open label, randomised, two-treatment, four-period, two-sequence, single-dose, crossover, fully replicated bioavailability study on Nitrofurantoin formulations comparing Nitrofurantoin 100 mg capsules of Ranbaxy Laboratories with Macrobid 100 mg capsules in healthy, adult, human subjects under fed conditions

DETAILED DESCRIPTION:
This was an open-label, randomized, single-dose, four period fully replicate crossover, relative bioavailability study performed on 40 healthy adult male and. A total of 35 completed the clinical phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range of 18-45 years.
* Be neither overweight nor underweight for his/her height as per the Life insurance Corporation of India height/weight chart for non-medical cases.
* Have voluntarily given written informed consent to participate in this study.
* Be of normal health as determined by medical history and physical examination of the subjects performed within 14 days prior to the commencement of the study.
* If female and:
* Of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or
* Is postmenopausal for at least I year; or
* Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* History of allergy to nitrofurantoin and/or other related drugs.
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Evidence of haemolysis (for glucose-6-phosphotase) deficiency.
* Presence of disease markers of HIV 1 and 2, Hepatitis B and C viruses or syphilis infection.
* Female volunteers demonstrating a positive pregnancy test.
* Female volunteers who are currently breastfeeding.
* Presence of values which are significantly different from normal reference ranges (as defined in Appendix 5) and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Positive for urinary screen testing of drugs of abuse (opiates and cannabinoids)
* Presence of values which are significantly different from normal reference ranges (as defined in Appendix 5) and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Clinically abnormal chemical and microscopic examination of udne defined as presence of RI3C, WBC (>4/HPF), epithelial cells (>4/HPF), glucose (positive) or protein (positive).
* Clinically abnormal ECG or Chest X-ray. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes, glaucoma or gout.
* History of any psychiatric illness which may impair the ability to provide written informed consent.
* Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unify.equivalent to half pint of beer or ! glass of wine or 1 measure of spirit)or have difficulty in abstaining for the duration of each study period.
* Use of any enzyme modi~ing drugs within 30 days prior to Day 1 of this study.
* Participation in any clinical trial within 12 weeks preceding Day ! of this study.
* A haemoglobin concentration of less than 7 % of lower limit of reference range e.g. 13 gm % for reference range of 14-18 gm at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09; Primary Completion 2003-10 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Research Laboratories, Gurgaon, Haryana, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html